CLINICAL TRIAL: NCT00518024
Title: Safety and Effectiveness of Bilateral Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation) in the Treatment of Chronic Tinnitus
Brief Title: Safety and Effectiveness of Repetitive Transcranial Magnetic Stimulation in the Treatment of Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other); CenTrial GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PL 525/1-1
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Tinnitus
Keywords: tinnitus; transcranial magnetic stimulation; treatment; cortex
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Bilateral theta burst stimulation to the secondary auditory cortex
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- 2 (Experimental): Bilateral theta burst stimulation to the tertiary auditory cortex
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- 3 (Sham Comparator): Bilateral theta burst stimulation to a non-cortical region
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS) — Bilateral Theta Burst Stimulation

SUMMARY:
Tinnitus, i.e., the perception of sounds or noise in the absence of auditory stimuli, is a frequent and often severely disabling symptom of different disorders of the auditory system. There are currently no causal treatments. Using repetitive transcranial magnetic stimulation (rTMS), we have previously demonstrated that the temporoparietal cortex is critically involved in tinnitus perception and that tinnitus can be reduced by rTMS applied to these cortical regions. Therefore, it is reasonable to test rTMS as a potential new treatment strategy against tinnitus. At this stage, small pilot studies indicate some effect on tinnitus impairment but the reduction is predominantly reported to be transient, with high interindividual variability, and questionable clinical relevance. Moreover, the optimal stimulation area is unclear.

Here, we use theta burst stimulation (TBS), a new rTMS paradigm for the prolonged modulation of cortical activity. The aim of this study is to test safety and effectivity of 4 weeks of daily bilateral TBS to two cortical areas on chronic tinnitus compared to sham-stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjective tinnitus > 6 mo , < 5 ys

Exclusion Criteria:

* Objective tinnitus
* Seizures
* Brain trauma
* Brain surgery
* Pacemaker
* intake of: benzodiazepines, antiepileptics, neuroleptics
* Suicidality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)

PRIMARY OUTCOMES:
Tinnitus severity (Tinnitus Questionnaire) | after the end of treatment

SECONDARY OUTCOMES:
Visual Analog Scale (Tinnitus Loudness); Visual Analog Scale (Tinnitus Annoyance); Visual Analog Scale (Tinnitus Change); Becks Depression Inventory; Symptom Check List; Audiogram; Speech Audiometry | after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, M.D., Principal Investigator — University of Tuebingen, Department of General Psychiatry
Locations (1):
- Department of General Psychiatry, University Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Background] Plewnia C, Reimold M, Najib A, Reischl G, Plontke SK, Gerloff C. Moderate therapeutic efficacy of positron emission tomography-navigated repetitive transcranial magnetic stimulation for chronic tinnitus: a randomised, controlled pilot study. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):152-6. doi: 10.1136/jnnp.2006.095612. Epub 2006 Aug 4. PMID 16891384
- [Background] Plewnia C, Reimold M, Najib A, Brehm B, Reischl G, Plontke SK, Gerloff C. Dose-dependent attenuation of auditory phantom perception (tinnitus) by PET-guided repetitive transcranial magnetic stimulation. Hum Brain Mapp. 2007 Mar;28(3):238-46. doi: 10.1002/hbm.20270. PMID 16773635
- [Background] Smith JA, Mennemeier M, Bartel T, Chelette KC, Kimbrell T, Triggs W, Dornhoffer JL. Repetitive transcranial magnetic stimulation for tinnitus: a pilot study. Laryngoscope. 2007 Mar;117(3):529-34. doi: 10.1097/MLG.0b013e31802f4154. PMID 17334317
- [Background] Rossi S, De Capua A, Ulivelli M, Bartalini S, Falzarano V, Filippone G, Passero S. Effects of repetitive transcranial magnetic stimulation on chronic tinnitus: a randomised, crossover, double blind, placebo controlled study. J Neurol Neurosurg Psychiatry. 2007 Aug;78(8):857-63. doi: 10.1136/jnnp.2006.105007. Epub 2007 Feb 21. PMID 17314192
- [Background] Fregni F, Marcondes R, Boggio PS, Marcolin MA, Rigonatti SP, Sanchez TG, Nitsche MA, Pascual-Leone A. Transient tinnitus suppression induced by repetitive transcranial magnetic stimulation and transcranial direct current stimulation. Eur J Neurol. 2006 Sep;13(9):996-1001. doi: 10.1111/j.1468-1331.2006.01414.x. PMID 16930367
- [Background] De Ridder D, Verstraeten E, Van der Kelen K, De Mulder G, Sunaert S, Verlooy J, Van de Heyning P, Moller A. Transcranial magnetic stimulation for tinnitus: influence of tinnitus duration on stimulation parameter choice and maximal tinnitus suppression. Otol Neurotol. 2005 Jul;26(4):616-9. doi: 10.1097/01.mao.0000178146.91139.3c. PMID 16015156
- [Background] Kleinjung T, Eichhammer P, Langguth B, Jacob P, Marienhagen J, Hajak G, Wolf SR, Strutz J. Long-term effects of repetitive transcranial magnetic stimulation (rTMS) in patients with chronic tinnitus. Otolaryngol Head Neck Surg. 2005 Apr;132(4):566-9. doi: 10.1016/j.otohns.2004.09.134. PMID 15806046
- [Background] Eichhammer P, Langguth B, Marienhagen J, Kleinjung T, Hajak G. Neuronavigated repetitive transcranial magnetic stimulation in patients with tinnitus: a short case series. Biol Psychiatry. 2003 Oct 15;54(8):862-5. doi: 10.1016/s0006-3223(02)01896-6. PMID 14550687
- [Background] Plewnia C, Bartels M, Gerloff C. Transient suppression of tinnitus by transcranial magnetic stimulation. Ann Neurol. 2003 Feb;53(2):263-6. doi: 10.1002/ana.10468. PMID 12557296
- [Derived] Arfeller C, Vonthein R, Plontke SK, Plewnia C. Efficacy and safety of bilateral continuous theta burst stimulation (cTBS) for the treatment of chronic tinnitus: design of a three-armed randomized controlled trial. Trials. 2009 Aug 21;10:74. doi: 10.1186/1745-6215-10-74. PMID 19698089